CLINICAL TRIAL: NCT02184975
Title: Randomized Clinical Trial Comparing Cold Knife Conization of the Cervix With and Without Lateral Hemostatic Sutures
Brief Title: Cold Knife Conization With and Without Lateral Hemostatic Sutures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ricardo dos Reis, Medical doctor, Barretos Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Conization1
Record Dates: First submitted 2014-06-20; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervix Neoplasms
Keywords: cold knife conization; lateral hemostatic sutures; cervix
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Conization; Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stitches (Experimental): Cold Knife Conization with stitches
  Interventions: Procedure: Cold Knife Conization with stitches
- No stitches (Active Comparator): Cold Knife Conization without stitches
  Interventions: Procedure: Cold knife Conization without stitches

INTERVENTIONS:
Procedure: Cold Knife Conization with stitches — In the research arm patients who underwent cold-knife conization of the cervix underwent hemostatic sutures laterally to the cervix, at localization of 3 and 9 hours with 2-0 vicryl thread. These sutures were held prior to the onset of cold conization of the cervix.
  Other Names: Cold Knife conization with sutures; Cervix hemostatic sutures
  Arms: Stitches
Procedure: Cold knife Conization without stitches — In the research arm patients who underwent cold-knife conization of the cervix have not undergone hemostatic sutures laterally to the cervix, at localization of 3 and 9 hours with 2-0 vicryl thread. After patient anesthesia and routine antisepsis was performed, cold knife conization of the cervix was performed.
  Other Names: Cervix conization without hemostatic sutures; Cold knife conization without lateral sutures
  Arms: No stitches

SUMMARY:
The treatment of high grade Cervical Intraepithelial Neoplasia (CIN) 2, 3 is defined according to the colposcopic evaluation of the patient. In case colposcopy findings are satisfactory (visible squamocolumnar junction), both ablative and excisional methods are adequate. In the middle of the 20th century, lateral hemostatic sutures were added to the cold knife conization surgical technique to reduce blood loss. Some authors recommend that these branches should be ligated, but it remains unclear whether these sutures are actually effective in reducing bleeding.This study compared blood loss during cold knife conization of the cervix with and without lateral hemostatic sutures.

DETAILED DESCRIPTION:
This is a study that will evaluate two groups of patients undergoing cold-knife conization for cervical intraepithelial neoplasia high grade where 50% will undergo hemostatic sutures in the lateral cervical and 50% of patients will not be subjected to these sutures. The main objective of the study is to evaluate the amount of intraoperative bleeding.

ELIGIBILITY:
Inclusion Criteria:

* indication of cold knife conization

Exclusion Criteria:

* conization using techniques other than the cold knife;
* previous cervical conization using any other technique;
* previous pelvic radiotherapy;
* pregnancy; and
* refusal to participate in the study

Ages: 15 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Intraoperatory vaginal bleeding | Intraoperatory
  The intraoperatory bleeding will be measure by weigh the gauze in grams (g).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo D Reis, MD, Study Chair — Hospital de Clinicas de Porto Alegre-Brazil
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Bueno LR, Binda M, Monego H, Scherer RL, Rolim KM, Bottini AL, Fregnani JH, dos Reis R. Randomized clinical trial comparing cold knife conization of the cervix with and without lateral hemostatic sutures. Int J Surg. 2015 Jun;18:224-9. doi: 10.1016/j.ijsu.2015.04.081. Epub 2015 Apr 30. PMID 25937157